CLINICAL TRIAL: NCT01559103
Title: A Double-blind, Placebo-controlled, Randomized Study in Rheumatoid Arthritis Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of MEDI5117 (Anti-IL-6)
Brief Title: Study to Assess the Safety and Tolerability of MEDI5117 in Rheumatoid Arthritis Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NN6018-4789; 2011-005402-29 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Phase I; Biologic
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MEDI5117 (Experimental): Intravenous infusion administered over 60 minutes
  Interventions: Biological: MEDI5117
- MEDI5117 Placebo (Placebo Comparator): Intravenous infusion administered over 60 minutes
  Interventions: Biological: MEDI5117 Placebo

INTERVENTIONS:
Biological: MEDI5117 — Intravenous infusion administered over 60 minutes, will be one of the following doses: 30, 100, 300, or 600 mg
  Arms: MEDI5117
Biological: MEDI5117 Placebo — Intravenous infusion administered over 60 minutes
  Arms: MEDI5117 Placebo

SUMMARY:
Study to assess the safety and tolerability of MEDI5117 in Rheumatoid Arthritis patients

DETAILED DESCRIPTION:
A Double-blind, Placebo-controlled, Randomized Study in Rheumatoid Arthritis Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of MEDI5117 (anti-IL-6)

ELIGIBILITY:
Inclusion Criteria:

* Active Rheumatoid Arthritis (RA) for 6 months or more.
* Males or nonpregnant, nonlactating femails aged 20 to 75 years, inclusive.
* Body Mass Index (BMI) between 19 and 36 kg/m2 and weight between 50 and 145 kg, inclusive.
* Males, unless surgically sterile, must use 2 effective methods of birth control from Day 1 through follow-up.

Exclusion Criteria:

* History or presence of any clinically significant disease or disorder which has not been stable over the previous 3 months.
* History of liver disease, bilirubin elevations, or Gilbert's Syndrome.
* Any systematic inflammatory condition in addition to RA (polymyalgia rheumatica, giant cell arthritis, systemic lupus, gout, pyrophosphate arthropathy).
* Current, chronic pain disorders including fibromyalgia and chronic regional pain syndromes or chronic fatigue syndromes.
* Intramuscular steroid injection or intraarticular steroid injection within 1 month of enrollment.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-05-31 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2014-02-28 (Actual)

PRIMARY OUTCOMES:
Description of the safety profile in terms of adverse events, blood pressure, pulse, temperature, ECG (Electrocardiogram), physical examination, and safety laboratory variables. | From Baseline up to 64 weeks

SECONDARY OUTCOMES:
Description of pharmacokinetics in terms of Maximum serum concentration (Cmax), time to Cmax (tmax), terminal rate constant(λz), terminal half-life (t1/2 λz). | From Day 1 Predose, 2h, 12h, 24h, day 7, week 2, 3, 4, 6, 8, 12, 16, 20, 24, 32, 40, 48, 56 and week 64.
Description of pharmacokinetics in terms of area under the serum concentration-time curve from zero to the time of the last quantifiable concentration [AUC(0-t)] and from zero to infinity (AUC). | From Day 1 Predose, 2h, 12h, 24h, day 7, week 2, 3, 4, 6, 8, 12, 16, 20, 24, 32, 40, 48, 56 and week 64.
Description of pharmacokinetics in terms of area under the serum concentration-time curve from zero to the time of concentration at Weeks 6 and 12 [AUC(0-6w) and AUC(0 12w)]. | From Day 1 Predose, 2h, 12h, 24h, day 7, week 2, 3, 4, 6, 8, 12, 16, 20, 24, 32, 40, 48, 56 and week 64.
Descriptions of pharmacokinetics in terms of systemic clearance (CL), volume of distribution during terminal phase (Vz), and volume of distribution at steady state (Vdss). | From Day 1 Predose, 2h, 12h, 24h, day 7, week 2, 3, 4, 6, 8, 12, 16, 20, 24, 32, 40, 48, 56 and week 64.
Description of pharmacodynamics in terms of total interleukin 6 (IL-6) and free IL-6 (exploratory) in plasma and high sensitive C-reactive protein (hs-CRP) pre and post MEDI5117 or placebo administration and their corresponding change from baseline. | From Baseline day -1 to week 64
Description of immunogenicity in terms of positive or negative for the presence of antidrug antibodies against MEDI5117 in blood. | From Baseline day -1 to week 64

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (3):
- Novo Nordisk Investigational Site, Overland Park, Kansas, United States
- Novo Nordisk Investigational Site, Berlin, Germany
- Novo Nordisk Investigational Site, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com